CLINICAL TRIAL: NCT00936468
Title: Randomized, Double Blind, Controlled Phase II Trial of the Safety, Tolerability and Immunogenicity of Fluzone® Inactivated Trivalent Influenza Virus Vaccine Administered With and Without JVRS-100 Adjuvant in Subjects 65 Years and Older
Brief Title: Safety, Tolerability and Immunogenicity of Fluzone® With and Without JVRS-100 in Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colby Pharmaceutical Company (Industry)
Responsible Party: Maggie Sisti, Juvaris
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-100-002
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Influenza
Keywords: Elderly influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fluzone® vaccine with JVRS-100 (3.75ug) (Experimental): One vaccination on Day 0 with Fluzone® vaccine at 45 ug mixed with JVRS-100 adjuvant at 3.75ug given by IM injection to the upper deltoid.
  Interventions: Biological: Fluzone® vaccine with JVRS-100 adjuvant or Fluzone alone
- Fluzone® vaccine with JVRS-100 (7.5ug) (Experimental): One vaccination on Day 0 with Fluzone® vaccine at 45 ug mixed with JVRS-100 adjuvant at 7.5ug given by IM injection to the upper deltoid.
  Interventions: Biological: Fluzone® vaccine with JVRS-100 adjuvant or Fluzone alone
- Fluzone® vaccine with JVRS-100 (25ug) (Experimental): One vaccination on Day 0 with Fluzone® vaccine at 45 ug mixed with JVRS-100 adjuvant at 25ug given by IM injection to the upper deltoid.
  Interventions: Biological: Fluzone® vaccine with JVRS-100 adjuvant or Fluzone alone
- Fluzone® vaccine alone (Experimental): One vaccination on Day 0 with Fluzone vaccine at 45 ug given by IM injection in the upper deltoid.
  Interventions: Biological: Fluzone® vaccine with JVRS-100 adjuvant or Fluzone alone

INTERVENTIONS:
Biological: Fluzone® vaccine with JVRS-100 adjuvant or Fluzone alone — One vaccination on Day 0 of Fluzone® vaccine at 45ug mixed with one of three doses (3.75ug, 7.5ug, 25ug) of JVRS-100 adjuvant versus Fluzone® vaccine at 45ug alone.

SUMMARY:
This study is designed to determine the optimal dose of JVRS-100 and assess safety, tolerability and immunogenicity of Fluzone® vaccine administered with JVRS-100 adjuvant at one of three dose levels compared to Fluzone® vaccine administered alone, in 472 adults aged ≥65 years.

DETAILED DESCRIPTION:
Approximately 472 subjects will be enrolled in this study. The study population will include elderly male and female subjects aged ≥65 years who are living in the community (including assisted living environments) and who are very fit to moderately frail.

One hundred subjects (approximately 25 in each treatment arms) will be vaccinated, and 14 days will elapse during which safety parameters are monitored by a Data and Safety Monitoring Board (DSMB), before randomizing the remaining 372 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Be adult volunteers aged ≥65 years
* Live in the community, independently or in an assisted living environment
* Be Class 1-5, as defined by the CSHA-CFS
* If female, will be post-menopausal
* Will be available for the duration of the trial (21-day On Study Period) and Follow-Up (4 and 9 months after vaccination)
* Be 'probably not demented' on the Mini-Cog test
* Provide informed consent
* Agree to defer receipt of vaccination of novel H1N1 (swine) influenza until after completion of the Day 28 study procedures

Exclusion Criteria:

* Known allergy to eggs or other components of the vaccine.
* History of severe reaction of any kind to conventional influenza vaccines
* Be Class 6-7 in the CSHA-CFS or be institutionalized (e.g., in a nursing home)
* Requiring nursing home-level equivalent care at home or within a community assisted living environment
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine.
* Significant cardiovascular disease (e.g., NYHA class 3 through 4 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled ventricular cardiac arrhythmias); resting heart rate >100;
* A history of chronic obstructive pulmonary disease or history of other lung disease requiring chronic steroid treatment in excess of a bioequivalent dose of 10 mg prednisone daily; a combined history of lung disease and anemia.
* Evidence of significant (more than 10 pounds) of unintentional weight loss in the last year.
* Changed residence or become hospitalized in the last 6 months.
* Combined history of depression and anemia.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Use of any investigational product within 60 days preceding the administration of the study vaccine, or planned use during the study period.
* Seropositive to HIV or HCV or positive for HBsAg
* Body temperature >38.1°C (100.6°F) or acute illness within 3 days prior to vaccination (subject may be rescheduled)
* History of excessive alcohol consumption, drug abuse, or significant psychiatric illness.
* Be 'probably demented' on the Min-Cog test
* Need for guardian assistance in completing informed consent
* Has received vaccination for novel H1N1 (swine) influenza

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 472 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety: The primary safety endpoint of this trial will be the evaluation of adverse events incidence rates between treatment groups. | Active Study Duration
Immunogenicity: Dose-response analysis of HAI geometric mean titers (GMT) | Day 0, 21, 28, Month 4 and 9

SECONDARY OUTCOMES:
Safety: Comparison of AE rates at intervals between treatment groups. | Active Study Duration
Immunogenicity: Comparison of Fluzone® with JVRS-100 by examining seroprotection and seroconversion rates to various antigens, duration of HAI antibody titers, and assessment of cross-reactive HAI responses against drifted strains. | Day 0, 21, 28 and Month 4 and 9
T-cell responses will be measured. | Day 0, 7, 14 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sheldon, MD, Principal Investigator — Miami Research Associates, FL; Casey Johnson, DO, Principal Investigator — Johnson County Clin-Trials, KS; Stephan Sharp, MD, Principal Investigator — Clinical Research Associates, TN; Aurora Pop-Vicas, MD, Principal Investigator — Memorial Hospital, RI; James Borders, MD, Principal Investigator — Central Kentucky Research Associates, KY; Rex Biedenbender, MD, Principal Investigator — Eastern Virginia Medical School, VA; Derek Muse, M.D., Principal Investigator — Jean Brown Research